CLINICAL TRIAL: NCT05853770
Title: Effects of School-Based TGfU Volleyball Intervention on Physical Fitness and Body Composition in Primary School Students: A Cluster-Randomized Trial
Brief Title: Effects of Volleyball Intervention on Health-related Fitness in Primary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nis (Other)
Collaborators: University of Milan (Other); University of Ljubljana (Other); University of Banja Luka (Other)
Responsible Party: Principal Investigator, Darko Stojanovic, Assistant Professor, University of Nis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04-2100
Record Dates: First submitted 2023-04-20; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Physical Inactivity; Adolescent Obesity; Physical Fitness; Body Composition; Healthy Lifestyle; Exercise
Keywords: physical activity; exercise training; physical education; volleyball; small-sided games; health-related fitness; body composition; physical fitness; adolescents; primary school
MeSH Terms: conditions — Sedentary Behavior; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGfU volleyball intervention (Experimental): According to the national curriculum, children in Serbia must attend three regular physical education (PE) classes per week.
  Besides attending two regular PE classes, participants in the experimental group also followed a 16-week TGfU volleyball intervention that was implemented during the third PE class. The total number of sessions: 32 regular PE + 16 TGfU volleyball intervention .
  Interventions: Other: TGfU volleyball intervention
- Control group (Active Comparator): Control group (CG) participants followed the national physical education curriculum. The CG participants conducted three regular PE classes per week or 48 regular PE classes in total.
  Interventions: Other: Regular physical education classes

INTERVENTIONS:
Other: TGfU volleyball intervention — Duration of intervention: 16 week; Duration of each session: 45 minutes; Frequency: One session per week during the third PE class;
  The structure of each TGfU session had three parts:
  The introduction part comprised 10 minutes of moderate-intensity warm-up activities; The main part comprised mini-volleyball and small-sided games (25-30 minutes); The last part of the session was the cool-down period (5 min).
  Arms: TGfU volleyball intervention
Other: Regular physical education classes — Regular physical education classes following national physical education curriculum for second semester of seventh grade in primary school in Serbia.
  Arms: Control group

SUMMARY:
The goal of this study is to find out if doing a 16-week volleyball program integrated in physical education classes at school can make primary school students stronger, faster, and have better endurance. The study also wants to see whether the program can lead to changes in the students' body weight, body fat, and muscle mass.

DETAILED DESCRIPTION:
Eighty-eight healthy primary school students (mean age 13.3 years) were randomized to a TGfU volleyball intervention group (VG) or a control group (CG). CG participants attended three regular physical education (PE) classes per week, while VG participants attended two regular PE classes and a TGfU volleyball intervention that was implemented in the third PE class. The main part of each volleyball intervention session was based on the "Teaching Games for Understanding" (TGfU) model. This approach emphasizes the development of fundamental skills and tactical understanding of the game by utilizing modified games, such as small-sided games and mini-volleyball. By using this method, participants are able to increase their interaction with the ball and engage in moderate-to-vigorous gameplay intensity more frequently. The primary study outcomes were assessed before and after the 16-week intervention for both VG and CG participants. The main hypothesis is that implementation of the TGfU volleyball intervention in the physical education curriculum will lead to greater improvement in body composition and physical fitness outcomes among seventh-grade primary school students compared to those who receive traditional physical education classes, demonstrating that this intervention can be an effective method for reducing adiposity and promoting physical fitness levels among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* seventh grade primary school students
* were not exempt from participating in physical education classes
* did not have any health conditions (pediatric disease, orthopedic conditions, injuries, respiratory or cardiovascular disease)
* voluntary participation
* obtained informed consent from parents or legal guardians

Exclusion Criteria:

* exempted from participating in physical education classes
* currently participating in other interventions
* the presence of acute or chronic infectious disease
* the presence of injury
* not able to attend all intervention sessions
* not obtaining informed consent from parents or legal guardians
* do not want to participate voluntary

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-02-04 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | Baseline, after 16 weeks
  Cardiorespiratory fitness is considered one of the most powerful health-related markers in adolescents. In this study, cardiorespiratory fitness is assessed using the 20-m shuttle-run test, which was adopted from the Eurofit test battery. Scoring is obtained as VO2max values (mL/kg/min).

SECONDARY OUTCOMES:
Change in Flexibility | Baseline, after 16 weeks
  Sit-and-Reach test is used for flexibility assessment. Measurements are recorded to the nearest centimeter.
Change in Speed | Baseline, after 16 weeks
  Sprinting abilities are assessed through a 30 m sprint test. Sprinting times are recorded with an accuracy of 0.01 seconds.
Change in Strength | Baseline, after 16 weeks
  Lower limb explosive strength is assessed through vertical jump tests, squat and countermovement jumps. Jump heights were recorded to the nearest centimeter.
Change in Agility | Baseline, after 16 weeks
  Agility is assessed utilizing Agility T-test. Time taken to finish the test was recorded with an accuracy of 0.01 seconds.
Change in Body Fat Percentage | Baseline, after 16 weeks
  Total body fat percentage assessed using bioelectric impendence method.
Change in Body Weight | Baseline, after 16 weeks
  Body Weight assessed using digital scale and recorded in kilograms.
Change in BMI | Baseline, after 16 weeks
  Body Mass Index (BMI) is calculated by dividing a person's weight in kilograms by the square of their height in meters. BMI = weight (kg) / height^2 (m^2).
Change in Muscle Mass Percentage | Baseline, after 16 weeks
  Total muscle mass percentage in body, assessed using bioelectric impendence method.
Change in Sum of skinfolds | Baseline, after 16 weeks
  Measurements of skinfold thicknesses were obtained using calibrated caliper at five skinfold sites calf, suprailiac, subscapular, triceps, and biceps (recorded in mm). The sum of skinfolds was calculated by summing the thicknesses of all five skinfold sites.

CONTACTS AND LOCATIONS:
Overall Officials: Toplica Stojanovic, Study Chair — University of Banja Luka
Locations (1):
- Primary School "Dušan Radović", Niš, Serbia

IPD SHARING:
Plan to Share IPD: No